CLINICAL TRIAL: NCT01331616
Title: A Prospective Single Institution Study of Optic Neuropathy in 10 Patients With Glioblastoma Receiving Bevacizumab
Brief Title: Optic Neuropathy in 10 Patients With Glioblastoma Receiving Bevacizumab
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Sponsor: West Penn Allegheny Health System (Other)
Responsible Party: Principal Investigator, Dawnmarie DeFazio, Physician, West Penn Allegheny Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC-5148
Record Dates: First submitted 2011-04-01; First posted 2011-04-08 (Estimated); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Glioblastoma; Optic Neuropathy
Keywords: Prospective study; Glioblastoma; Avastin; Visual Evoked Potential; Optic neuropathy; Chemo-radiotherapy
MeSH Terms: conditions — Glioblastoma; Optic Nerve Diseases | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab (Avastin) (Experimental)
  Interventions: Drug: Bevacizumab (Avastin)

INTERVENTIONS:
Drug: Bevacizumab (Avastin) — Dosage is: 10 mg/kg every 2 weeks as monotherapy or in combination (unlabeled) with irinotecan. Patients will also receive Radiotherapy prior to beginning chemotherapy.

SUMMARY:
Does treatment with bevacizumab (Avastin) in combination with prior or current radiotherapy lead to optic neuropathy?

DETAILED DESCRIPTION:
The investigators research will focus on patients prior to them beginning treatment with bevacizumab (Avastin), by undergoing a baseline visual examination with Visual evoked Potentials testing. This will allow testing of the patient's optic nerve function bilaterally. Patients will then begin their normally scheduled treatment with avastin, and other chemotherapeutic agents, as well any radiation treatments scheduled. Once patients have completed their treatment with avastin for 6-8 weeks, they will then undergo their second Visual Evoked Potential testing, with both studies then being compared for any changes within the optic nerves. Patients will also be recommended to have stringent follow up with an Ophthalmologist to include confrontational visual field testing, external and anterior segment examination, and dilated fundus examination. The investigators main objective is to assess whether or not bevacizumab causes a direct toxic effect on patient's optic nerves leading to an acute/subacute optic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed w Glioblastoma grade IV, and scheduled to begin chemo radiotherapy with Avastin

Exclusion Criteria:

* No diagnosis of GBM, not scheduled to begin treatment with avastin in combination with radiotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Measurement of Visual Evoked Potentials (optic nerve function and visual processing) and optic nerve function in 10 patients. | 1 year
  Does Avastin lead to optic neuropathy in combination w chemo-radiotherapy? Our research will focus on patients prior to them beginning treatment with bevacizumab (Avastin), by undergoing Visual evoked Potentials testing. This will allow testing of the patient's optic nerve function bilaterally. In our study of VEP, we will be measuring optic nerve function, to asses if there has been any damage.

SECONDARY OUTCOMES:
Number of patients diagnosed with optic neuropathy following treatment with chemo and radiation in combination with avastin treatment | 1 year
  The investigators will compare the results of the patient's Visual Evoked Potential (VEP) testing performed prior to treatment with Avastin and chemo-radiotherapy to the results of the VEP after completion to assess optic nerve function; and any signs of direct optic neuropathy In our study the investigators will compare the results of the Visual Evoked Potential results performed prior to the chemoradiation to results of the Visual Evoked Potential after completion of standard-of-care treatment for glioblastoma.